CLINICAL TRIAL: NCT02712424
Title: A Phase 2, Randomized, Placebo-Controlled, Double-Blind, Study of the Prevention of Infection With Mycobacterium Tuberculosis Among Adolescents Who Have Previously Received BCG
Brief Title: DAR-901 TB Booster Vaccine to Prevent TB in Adolescents
Acronym: DAR-PIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, C. Fordham von Reyn, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 29001
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Tuberculosis
Keywords: Vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAR-901 (Active Comparator): 0.1 mL intradermal injection of 1 mg DAR-901
  Interventions: Biological: DAR-901
- Placebo (Placebo Comparator): 0.1 mL intradermal injection of sterile saline for human use
  Interventions: Biological: Sterile saline placebo

INTERVENTIONS:
Biological: DAR-901
  Arms: DAR-901
Biological: Sterile saline placebo
  Arms: Placebo

SUMMARY:
DAR-901 booster vaccine or placebo will be administered to adolescents in Tanzania primed with BCG to determine if immunization reduces the risk of TB infection

DETAILED DESCRIPTION:
DAR-901 whole cell booster vaccine to prevent TB infection in adolescents ("DAR-PIA")

This is a Phase II, 3-injection, randomized, controlled trial of DAR-901 to be conducted in 13-15 year old adolescents in Tanzania previously immunized with BCG. DAR-901 is a whole cell inactivated non-tuberculous mycobacterial vaccine manufactured from the Master Cell Bank of SRL-172 that was used in the successful Phase III DarDar Trial in Tanzania. The goals are to establish the safety and efficacy of DAR-901 in preventing infection with TB. The 1 mg dose was selected during the current Phase I dose-escalation trial of DAR-901 in the US being conducted by Dartmouth and Aeras. The 1 mg dose corresponds to the dose of SRL 172 used in the DarDar Trial.

All subjects will be screened by the T-spot® IGRA (Oxford Immunotec, Oxford, England) for evidence of TB infection. All screened subjects will have a structured interview to identify risk factors for TB infection (=positive IGRA). IGRA-positive subjects will be referred for further evaluation and will not be entered in the immunization phase of the trial.

It is estimated that 1000 adolescents will need to be screened to identify a total of 650 IGRA-negative adolescents in the immunization phase of the trial. Subjects will be and randomized 1:1 to DAR-901 or saline control at 0, 2 and 4 months. Doses will be administered by intradermal (ID) injection in the deltoid area. IGRA testing will be repeated before dose 2, at 14 months, and again at 24 months.

This three year study began in the first quarter of 2016 in Dar es Salaam, is funded by GHIT-Japan and will be directed by Geisel School of Medicine at Dartmouth (PI, F. von Reyn) with collaborators at Muhimbili University of Health and Allied Sciences (MUHAS) in Tanzania and Tokyo Medical and Dental University in Japan.

ELIGIBILITY:
Inclusion Criteria: Negative IGRA at baseline -

Exclusion Criteria: Pregnancy, serious underlying disease

-

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 625 (Actual)
Dates: Start 2016-03; Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C Fordham von Reyn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Munseri P, Said J, Amour M, Magohe A, Matee M, Rees CA, Mackenzie T, Tvaroha S, Bailey-Kellogg C, Maro I, Wieland-Alter W, Adams LV, Horsburgh CR, Nakamura K, Arbeit RD, Pallangyo K, von Reyn CF. DAR-901 vaccine for the prevention of infection with Mycobacterium tuberculosis among BCG-immunized adolescents in Tanzania: A randomized controlled, double-blind phase 2b trial. Vaccine. 2020 Oct 27;38(46):7239-7245. doi: 10.1016/j.vaccine.2020.09.055. Epub 2020 Sep 29. PMID 33004239
- [Derived] Rees CA, Pineros DB, Amour M, Munseri P, Said J, Magohe A, Matee M, Pallangyo K, von Reyn CF. The potential of CBC-derived ratios (monocyte-to-lymphocyte, neutrophil-to-lymphocyte, and platelet-to-lymphocyte) to predict or diagnose incident TB infection in Tanzanian adolescents. BMC Infect Dis. 2020 Aug 18;20(1):609. doi: 10.1186/s12879-020-05331-w. PMID 32811463

RESULTS

PARTICIPANT FLOW:
Groups:
- DAR-901: 0.1 mL intradermal injection of 1 mg DAR-901
  DAR-901
- Placebo: 0.1 mL intradermal injection of sterile saline for human use
  Sterile saline placebo
Period: Overall Study
Arm/Group | DAR-901 | Placebo
Started | 315 | 310
Completed | 281 | 278
Not Completed | 34 | 32
Not completed — Lost to Follow-up | 34 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DAR-901 | Placebo | Total
Number analyzed (Participants) | 315 | 310 | 625
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 315 | 310 | 625
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (0.76) | 14.2 (0.75) | 14.15 (.755)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 169 | 361
  Male | 123 | 141 | 264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 315 | 310 | 625
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 315 | 310 | 625
IGRA negative [Count of Participants; unit: Participants] | 315 | 310 | 625

OUTCOME MEASURES:

1. Primary Outcome: New Infection With Mycobacterium Tuberculosis
Description: New infection with TB is based on conversion of IGRA
Time Frame: 3 years
Population: Conversion from IGRA neg to pos
Measure: Count of Participants; unit: Participants
Arm/Group | DAR-901 | Placebo
Number analyzed (Participants) | 315 | 310
Participants | 19 | 18

2. Secondary Outcome: Persistent New Infection With M. Tuberculosis
Description: New positive IGRA that is also positive on repeat ≥3 mos later
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | DAR-901 | Placebo
Number analyzed (Participants) | 315 | 310
participants | 10 | 5

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | DAR-901 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/310
Serious Adverse Events (participants affected / at risk) | 6/315 | 3/310
Other Adverse Events (participants affected / at risk) | 126/315 | 142/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAR-901 (N=315) | Placebo (N=310)
Tuberculosis (Infections and infestations) | 3 (3) | 2 (2) — Active TB was defined as an SAE for purpose of this study
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
HIV infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAR-901 (N=315) | Placebo (N=310)
Infections and infestations (Infections and infestations) | 73 (73) | 69 (310)
Other (General disorders) | 53 (53) | 73 (73)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02712424/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT02712424/SAP_001.pdf